CLINICAL TRIAL: NCT01026519
Title: A Single-dose, Double-Blind, Placebo-Controlled, Parallel Group Safety, Tolerability and Pharmacodynamic Study of Subcutaneous REGN88 in Subjects With Rheumatoid Arthritis Receiving Concomitant Methotrexate
Brief Title: A Safety and Tolerability Study of REGN88(SAR153191) in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6R88-RA-0803
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Dose 1 (Experimental): Active dose
  Interventions: Drug: REGN88
- Dose 2 (Experimental): Active dose
  Interventions: Drug: REGN88
- Dose 3 (Experimental): Active 3
  Interventions: Drug: REGN88
- Dose 4 (Placebo Comparator): Placebo dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: REGN88 — Single dose of REGN88 and 43 day follow up.
  Arms: Dose 1; Dose 2; Dose 3
Other: Placebo — Placebo to match REGN88 administration
  Arms: Dose 4

SUMMARY:
This is a single-dose, double-blind, placebo-controlled, parallel group safety, tolerability and pharmacodynamic study of subcutaneously (SC) administered REGN88 in rheumatoid arthritis patients who are receiving concomitant methotrexate. Four (4) parallel groups of 8 subjects each with active rheumatoid arthritis will be dosed SC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Subjects must weigh >50 and <100 kg
3. Diagnosis of Rheumatoid Arthritis (RA) as defined by the 1987 revised American College of Rheumatology (ACR) criteria with disease duration of no less than 6 months and ACR class I-III

Exclusion Criteria:

1. A history of Listeriosis or active tuberculosis (TB)
2. Persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the Screening Visit
3. History of prior articular or prosthetic joint infection
4. History of a hypersensitivity reaction, other than localized injection site reaction (ISR), to any biological molecule
5. Significant concomitant illness such as, but not limited to cardiac, renal, neurological, endocrinological, metabolic or lymphatic disease that would adversely affect the subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
hs-C reactive protein (hs-CRP) | 43 Days

SECONDARY OUTCOMES:
Subject's Assessment of Pain and Subject's Global Assessment of Disease activity | 43 Days

CONTACTS AND LOCATIONS:
Overall Officials: Allen Radin, MD, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Institute of Rheumatology under the Russian Academy of Medical Sciences, Moscow, Russia